CLINICAL TRIAL: NCT00531999
Title: An Open Label Study of the Impact on Insulin Sensitivity, Lipid Profile and Vascular Inflammation by Treatment With Lopinavir / Ritonavir (400 / 100 mg Twice Daily) or Raltegravir 400 mg Twice Daily in HIV Negative Male Volunteers.
Brief Title: Raltegravir Insulin Sensitivity Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St Stephens Aids Trust (Other)
Responsible Party: Dr Graeme Moyle, St Stephen's AIDS Trust
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: SSAT023
Record Dates: First submitted 2007-09-18; First posted 2007-09-19 (Estimated); Last update posted 2010-08-16 (Estimated); Status verified 2010-08

CONDITIONS: HIV Infections
Keywords: Raltegravir; Euglycaemic clamp; healthy volunteer
MeSH Terms: conditions — HIV Infections | interventions — Ritonavir; Lopinavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Raltegravir 400 mg twice daily for the first 14 days of the study. Lopinavir/ritonavir 400/100 mg twice daily for the last 14 days of the study
  Interventions: Drug: Raltegravir then lopinavir/ritonavir
- 2 (Active Comparator): * Lopinavir/ritonavir 400/100 mg twice daily for the first 14 days of the study.
  * Raltegravir 400 mg twice daily for the last 14 days of the study.
  Interventions: Drug: Lopinavir/ritonavir then raltegravir

INTERVENTIONS:
Drug: Raltegravir then lopinavir/ritonavir — raltegravir 400mg twice daily for first 14 days of study lopinavir/ritonavir 400/100mg twice daily for last 14 days of study
  Arms: 1
Drug: Lopinavir/ritonavir then raltegravir — lopinavir/ritonavir 400 mg twice daily for the first 14 days of the study raltegravir 400mg twice daily for the last 14 days of the study
  Arms: 2

SUMMARY:
The purpose of the study is to look at the effects of two different HIV medications on the body's response to insulin (a hormone that regulates blood sugar levels). This will be done using a method called the 'euglycaemic clamp'

The study will also investigate the effects of these drugs on blood fats and on circulating markers in the blood stream related to blood vessels (vascular inflammation markers).

DETAILED DESCRIPTION:
Subjects will undergo four euglycaemic clamp procedures in order to determine the extent of glucose disposal. The first clamp will be performed prior to the commencement of the first study drug administration, the second one following two weeks of study drug, the third after a two week washout period, prior to commencement of second study drug administration and the fourth after two weeks of the second study drug

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have documented negative HIV serology by ELISA and P24 antigen
* Subjects must be clinically well males aged between 18 to 60 years
* Fasting blood glucose, total cholesterol and triglycerides within normal limits
* Hepatic transaminases (AST and ALT) ≤ 3 × upper limit of normal (ULN)
* Adequate hematologic function (absolute neutrophil count ≥ 1,000/mm3; platelets ≥ 50,000/mm3; hemoglobin ≥ 8.0 g/dL)
* Serum amylase ≤ 1.5 × ULN (subjects with serum amylase > 1.5 × ULN will remain eligible if pancreatic lipase is ≤ 1.5 × ULN)
* Sexually active males must use condoms during the course of the study
* Life expectancy ≥ 1 year
* Willing and able to provide informed consent

Exclusion Criteria:

* Subjects with a waist hip ratio > 0.97 or BMI > 28 kg/m2 will be excluded
* Acute or chronic hepatitis B infection (determined by positive hepatitis B surface antigen result at the screening visit)
* Acute or chronic hepatitis C infection (determined by positive hepatitis C antibody result at the screening visit)
* Other metabolic syndrome or disease process in the opinion of the investigator likely to cause marked disturbance in glucose and lipid homeostasis including hypertension
* Receiving on-going therapy with any of the following:

  * Metabolically active medications
  * Any lipid-lowering medication
  * Hormonal agents (oestrogens or androgens)
  * Glucocorticoids
  * Beta-blockers
  * Thiazide diuretics
  * Thyroid preparations
  * Psychotropic agents
  * Anabolic steroids
  * Megestrol acetate

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2007-10; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in insulin sensitivity by euglycaemic clamp method | 2 weeks

SECONDARY OUTCOMES:
Change from baseline in serum levels of fasting cholesterol, triglycerides | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Greame Moyle, Principal Investigator — Chelsea & Westminser Healthcare NHS Trust
Locations (1):
- St Stephens Centre, Chelsea & Westminster Hospital, London, United Kingdom